CLINICAL TRIAL: NCT00215449
Title: Study in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DL-059
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2009-01

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; formoterol; formoterol fumarate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the investigational drug in the treatment of COPD in comparison with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD
* Current or prior history of cigarette smoking

Exclusion Criteria:

* Medical diagnosis of asthma
* Chest x-ray (CXR) prior to Day 1 diagnostic of significant disease other than COPD
* Significant condition or disease other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690
Dates: Primary Completion 2005-12 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Measure of lung function

SECONDARY OUTCOMES:
Change in lung function, as well as vital signs
Physical Exam results, Adverse Event reporting, etc

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - Research Site, Bessemer, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tuscon, Arizona
  - Research Site, Buena Park, California
  - Research Site, Encinitas, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, San Diego, California
  - Research Site, Sepulveda, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bay Pines, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Hines, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Butte, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Springfield, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Larchmont, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Easton, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Donohue JF, Hanania NA, Fogarty C, Campbell SC, Rinehart M, Denis-Mize K. Long-term safety of nebulized formoterol: results of a twelve-month open-label clinical trial. Ther Adv Respir Dis. 2008 Aug;2(4):199-208. doi: 10.1177/1753465808093934. PMID 19124372